CLINICAL TRIAL: NCT00002781
Title: PROCEDURES FOR BNCT PHASE-I STUDY OF MELANOMA IN THE EXTREMITIES
Brief Title: Boron Neutron Capture Therapy in Treating Patients With Stage III Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beth Israel Deaconess Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064811; NEDH-961207015; NCI-V96-0907
Record Dates: First submitted 1999-11-01; First posted 2004-09-02 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2000-04

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — 4-boronophenylalanine-fructose

INTERVENTIONS:
Drug: boronophenylalanine-fructose complex

SUMMARY:
RATIONALE: Boron neutron capture therapy may selectively kill tumor cells without harming normal tissue.

PURPOSE: Phase I trial to study the effectiveness of boron neuron capture therapy in treating patients with stage III melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the maximum tolerated dose of neutron irradiation that can be given in combination with borophenylalanine-fructose complex (BPA-F) in patients with stage III melanoma. II. Evaluate the safety of this regimen. III. Evaluate tumor response to this regimen.

OUTLINE: This is a dose-finding study. Patients receive a test dose of borophenylalanine-fructose complex (BPA-F) for biodistribution studies and undergo punch biopses of tumor and normal tissue to measure B-10 concentration. Later, a treatment dose of BPA-F over 1 hour is followed by neutron irradiation. Groups of 3 patients receive escalated doses of neutron irradiation until the maximum tolerated dose is determined. Patients who complete protocol treatment and continue to meet the eligibility criteria may re-enter the study, provided at least 6 months has elapsed since the completion of prior therapy and the field boundary for the new irradiation site is seperated from the boundary of the previously irradiated site. Patients are followed monthly for 12 months, then every 3-6 months as needed.

PROJECTED ACCRUAL: Approximately 15 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven melanoma that is clinical stage III Estimated clinical tumor depth 1.0-6.0 cm from the epidermis Tumor surface diameter no greater than 10 cm Grossly evident cutaneous or subcutaneous tumor nodules are eligible for irradiation

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70%-100% Life expectancy: More than 3 months Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No history of phenylketonuria Negative serum pregnancy test required of fertile women Adequate contraception required of fertile women during and for 6 months after the study

PRIOR CONCURRENT THERAPY: No prior radiotherapy to the target area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 1996-04

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Busse, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Boston University School of Medicine, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts